CLINICAL TRIAL: NCT01756391
Title: Allergens in Inner-City Schools and Childhood Asthma
Acronym: SICAS-1
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Wanda Phipatanakul, Associate Professor of Pediatrics, Boston Children's Hospital
Other Study IDs: R01 AI 0739654
Record Dates: First submitted 2012-12-20; First posted 2012-12-25 (Estimated); Results first posted 2014-12-08 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Asthma
Keywords: pediatric; childhood; allergy
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Asthma is a disease that affects more than 12% of Americans under the age of 18 for over 14 million missed school days per year, and is the number one cause of school absences in America. Elementary school children spend 6 to 10 hours a day in school, and most of that time is spent in one classroom. The goals of this project are to provide an understanding of exposure risk factors specific to the classroom. This is critical, because the classroom environment could potentially be considered as an effective target for prevention of inner-city asthma morbidity by reducing exposures to many symptomatic children through an intervention in the school classrooms.

ELIGIBILITY:
Inclusion Criteria:

* Grades K-8 the school year following spring recruitment (Ages 4-15)
* Attend one of the schools in the fall where permission obtained for classroom sampling.
* Able to provide assent and parent/guardian able to provide informed consent Physician-Diagnosed asthma AND Wheezing in the previous 12 months

Exclusion Criteria:

* Significant pulmonary diseases other than asthma that might influence test results or pose risks (e.g., cystic fibrosis, sarcoidosis, bronchiectasis)
* Cardiovascular disease that requires daily medication
* Taking a beta blocker
* Active smoker
* Unable to follow through with study visit or complete study procedures

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: elementary school students with asthma
Sampling Method: Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2008-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital, Boston, Boston, Massachusetts, United States

REFERENCES:
- [Background] Phipatanakul W, Matsui E, Portnoy J, Williams PB, Barnes C, Kennedy K, Bernstein D, Blessing-Moore J, Cox L, Khan D, Lang D, Nicklas R, Oppenheimer J, Randolph C, Schuller D, Spector S, Tilles SA, Wallace D, Sublett J, Bernstein J, Grimes C, Miller JD, Seltzer J; Joint Task Force on Practice Parameters. Environmental assessment and exposure reduction of rodents: a practice parameter. Ann Allergy Asthma Immunol. 2012 Dec;109(6):375-87. doi: 10.1016/j.anai.2012.09.019. No abstract available. PMID 23176873
- [Background] Bartnikas LM, Sheehan WJ, Hoffman EB, Permaul P, Dioun AF, Friedlander J, Baxi SN, Schneider LC, Phipatanakul W. Predicting food challenge outcomes for baked milk: role of specific IgE and skin prick testing. Ann Allergy Asthma Immunol. 2012 Nov;109(5):309-313.e1. doi: 10.1016/j.anai.2012.07.026. Epub 2012 Aug 21. PMID 23062384
- [Background] Rao DR, Gaffin JM, Baxi SN, Sheehan WJ, Hoffman EB, Phipatanakul W. The utility of forced expiratory flow between 25% and 75% of vital capacity in predicting childhood asthma morbidity and severity. J Asthma. 2012 Aug;49(6):586-92. doi: 10.3109/02770903.2012.690481. Epub 2012 Jun 28. PMID 22742446
- [Background] Rao D, Phipatanakul W. Impact of environmental controls on childhood asthma. Curr Allergy Asthma Rep. 2011 Oct;11(5):414-20. doi: 10.1007/s11882-011-0206-7. PMID 21710109
- [Result] Permaul P, Hoffman E, Fu C, Sheehan W, Baxi S, Gaffin J, Lane J, Bailey A, King E, Chapman M, Gold D, Phipatanakul W. Allergens in urban schools and homes of children with asthma. Pediatr Allergy Immunol. 2012 Sep;23(6):543-9. doi: 10.1111/j.1399-3038.2012.01327.x. Epub 2012 Jun 6. PMID 22672325
- [Result] Sheehan WJ, Hoffman EB, Fu C, Baxi SN, Bailey A, King EM, Chapman MD, Lane JP, Gaffin JM, Permaul P, Gold DR, Phipatanakul W. Endotoxin exposure in inner-city schools and homes of children with asthma. Ann Allergy Asthma Immunol. 2012 Jun;108(6):418-22. doi: 10.1016/j.anai.2012.04.003. Epub 2012 Apr 26. PMID 22626594
- [Result] Phipatanakul W, Bailey A, Hoffman EB, Sheehan WJ, Lane JP, Baxi S, Rao D, Permaul P, Gaffin JM, Rogers CA, Muilenberg ML, Gold DR. The school inner-city asthma study: design, methods, and lessons learned. J Asthma. 2011 Dec;48(10):1007-14. doi: 10.3109/02770903.2011.624235. Epub 2011 Oct 20. PMID 22010992
- [Result] Baxi SN, Sheehan WJ, Gaffin JM, Yodying J, Panupattanapong S, Lane JP, Fu C, Hoffman EB, Gold DR, Phipatanakul W. Agreement between parent and student responses to an asthma and allergy questionnaire in a diverse, inner-city elementary school population. Ann Allergy Asthma Immunol. 2011 Oct;107(4):371-3. doi: 10.1016/j.anai.2011.08.007. No abstract available. PMID 21962100
- [Derived] Hauptman M, Gaffin JM, Petty CR, Sheehan WJ, Lai PS, Coull B, Gold DR, Phipatanakul W. Proximity to major roadways and asthma symptoms in the School Inner-City Asthma Study. J Allergy Clin Immunol. 2020 Jan;145(1):119-126.e4. doi: 10.1016/j.jaci.2019.08.038. Epub 2019 Sep 23. PMID 31557500
- [Derived] Baxi SN, Sheehan WJ, Sordillo JE, Muilenberg ML, Rogers CA, Gaffin JM, Permaul P, Lai PS, Louisias M, Petty CR, Fu C, Gold DR, Phipatanakul W. Association between fungal spore exposure in inner-city schools and asthma morbidity. Ann Allergy Asthma Immunol. 2019 Jun;122(6):610-615.e1. doi: 10.1016/j.anai.2019.03.011. Epub 2019 Mar 20. PMID 30904580
- [Derived] Lai PS, Sheehan WJ, Gaffin JM, Petty CR, Coull BA, Gold DR, Phipatanakul W. School Endotoxin Exposure and Asthma Morbidity in Inner-city Children. Chest. 2015 Nov;148(5):1251-1258. doi: 10.1378/chest.15-0098. PMID 26087201

RESULTS

PARTICIPANT FLOW:
Groups:
- Observational Cohort: students with asthma grades K-8 after the spring screening attending schools where permission for sampling obtained
Period: Overall Study
Arm/Group | Observational Cohort
Started | 351
Completed | 319
Not Completed | 32

BASELINE CHARACTERISTICS:
Arm/Group | Observational Cohort
Number analyzed (Participants) | 351
Age, Continuous [Mean (Full Range); unit: years] | 7.9 [4 to 13]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169
  Male | 182
Region of Enrollment [Number; unit: participants] — Students with asthma from participating schools
  participants
    United States | 351

OUTCOME MEASURES:

1. Secondary Outcome: Days of Slowed Activity Due to Asthma
Time Frame: 12 months
Reporting Status: Not Posted

2. Secondary Outcome: Days of Exercise-induced Symptoms
Time Frame: 12 months
Reporting Status: Not Posted

3. Secondary Outcome: Days of Cough Without an Upper Respiratory Infection
Time Frame: 12 months
Reporting Status: Not Posted

4. Secondary Outcome: Nights of Wakening Due to Asthma Symptoms
Time Frame: 12 months
Reporting Status: Not Posted

5. Secondary Outcome: Number of Hospitalizations
Time Frame: 12 months
Reporting Status: Not Posted

6. Secondary Outcome: Emergency Department Visits
Time Frame: 12 months
Reporting Status: Not Posted

7. Secondary Outcome: Emergency Department Visits
Time Frame: 12 months
Reporting Status: Not Posted

8. Secondary Outcome: Unscheduled Physician/Health Care Visits
Time Frame: 12 months
Reporting Status: Not Posted

9. Secondary Outcome: Prednisone Bursts
Time Frame: 12 months
Reporting Status: Not Posted

10. Secondary Outcome: FEV1/FVC
Time Frame: 12 months
Reporting Status: Not Posted

11. Secondary Outcome: FEV1 Percent Predicted
Time Frame: 12 months
Reporting Status: Not Posted

12. Secondary Outcome: Percent Change in FEV1 After Short-acting Beta Agonist
Time Frame: 12 months
Reporting Status: Not Posted

13. Secondary Outcome: Exhaled Nitric Oxide Levels
Time Frame: 12 months
Reporting Status: Not Posted

14. Primary Outcome: Maximum Symptom Days/14 Days
Description: Largest value among the following:
  Number of days with wheezing, tightness in the chest, or cough Number of nights with disturbed sleep as a result of asthma Number of days on which the child had to slow down or discontinue play activities because of asthma
Time Frame: 14 days
Population: Those with appropriate follow up and school/home allergen exposure data and allergy sensitization data
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Observational Cohort
Number analyzed (Participants) | 284
days | 2.7 (4)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Observational Cohort
Serious Adverse Events (participants affected / at risk) | 0/351
Other Adverse Events (participants affected / at risk) | 0/351

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No